CLINICAL TRIAL: NCT07263256
Title: Surgical Treatment of Complex Regional Pain Syndrome by Median Nerve Decompression and Lesion-Specific Correction: A Clinical Study
Brief Title: Median Nerve Decompression for Complex Regional Pain Syndrome: A Clinical Study
Acronym: CRPS-SURG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jitka Fricova (Other)
Collaborators: Charles University, Czech Republic (Other); Ministry of Health, Czech Republic (Other Government); General University Hospital, Prague (Other)
Responsible Party: Sponsor-Investigator, Jitka Fricova, Head of Pain Management Center,MD, PhD. Ass.prof., Charles University, Czech Republic
Organization: Charles University, Czech Republic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRPS-MND-2014-2023; MH CZ-DRO-VFN64165 (Other Grant/Funding Number: Ministry of Health of the Czech Republic)
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Complex Regional Pain Syndrome I (CRPS I); Nerve Entrapment Syndrome
Keywords: Complex Regional Pain Syndrome; CRPS Type I; Neuropathic Pain; Median Nerve Decompression; Peripheral Nerve Surgery; Upper Limb Pain; Nerve Entrapment; Chronic Pain; Hand Surgery
MeSH Terms: conditions — Complex Regional Pain Syndromes; Charcot-Marie-Tooth Disease; Reflex Sympathetic Dystrophy; Neuralgia; Nerve Compression Syndromes; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Group A: Lesion-specific correction Group B: Median nerve decompression
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A - Lesion-Specific Surgical Correction (Active Comparator): Surgical correction of identifiable structural pathology, including hardware impingement, neuroma, tendon adhesion, scar tethering, or other mechanical causes of CRPS.
  Interventions: Procedure: Lesion-Specific Surgical Correction
- Arm B - Median Nerve Decompression (Active Comparator): Open decompression of the median nerve performed in patients without identifiable lesions but with nocturnal neuropathic pain suggestive of median nerve irritation.
  Interventions: Procedure: Median Nerve Decompression

INTERVENTIONS:
Procedure: Lesion-Specific Surgical Correction — Surgical correction of identifiable structural pathology, including hardware impingement, neuroma, tendon adhesion, scar tethering, or other mechanical causes of complex regional pain syndrome of the upper limb.
  Arms: Arm A - Lesion-Specific Surgical Correction
Procedure: Median Nerve Decompression — Surgical correction of identifiable structural pathology, including hardware impingement, neuroma, tendon adhesion, scar tethering, or other mechanical causes of complex regional pain syndrome of the upper limb.
  Arms: Arm B - Median Nerve Decompression

SUMMARY:
This clinical study evaluates the effectiveness of surgical treatment in patients with upper-limb complex regional pain syndrome (CRPS) diagnosed according to the Budapest criteria. Seventy-four patients were assessed between 2014 and 2023. Patients with identifiable structural pathology underwent lesion-specific surgical correction, while those without detectable lesions but with neuropathic nocturnal pain underwent decompression of the median nerve. Pain intensity was measured using the visual analogue scale (VAS) preoperatively, at 10-12 days, and at three months. The study aims to determine the speed and magnitude of pain improvement after targeted surgical intervention.

DETAILED DESCRIPTION:
Complex regional pain syndrome (CRPS) is a multifactorial neuropathic pain disorder that can occur after trauma or surgery and is often resistant to conservative treatment. Increasing evidence suggests that in a subset of patients, peripheral mechanical factors contribute significantly to symptom generation. This prospective clinical study evaluated the outcomes of targeted surgical treatment in patients with CRPS of the upper limb who met the Budapest diagnostic criteria.

From 2014 to 2023, seventy-four patients were examined. Thirty-eight patients presented with identifiable structural pathology, such as hardware impingement, neuroma, tendon adhesion, or scar tethering, and underwent lesion-specific surgical correction. Thirty-six patients had no detectable structural lesion but reported nocturnal neuropathic pain suggestive of median nerve irritation; these patients underwent decompression of the median nerve. Pain intensity was measured using the visual analogue scale (VAS) before surgery, at suture removal (10-12 days), and at three months postoperatively.

Patients with identifiable mechanical pathology demonstrated substantial improvement, with an average 7.2-point VAS reduction after six months. Patients who underwent median nerve decompression showed rapid and marked pain reduction, improving by 7.1 points within 10-12 days and 8.6 points within three months. Acute CRPS cases improved more than chronic ones, indicating an early therapeutic window before central sensitization becomes dominant. Only one chronic case failed to improve. The results suggest that timely surgical assessment and correction of peripheral nerve or soft-tissue factors may lead to rapid and significant clinical recovery in selected CRPS patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Complex Regional Pain Syndrome (CRPS) according to Budapest criteria
* Age ≥ 18 years
* Persistent symptoms despite previous conservative treatment
* Ability to understand the study information and provide informed consent
* Ability to adhere to postoperative follow-up

Exclusion Criteria:

* Active local or systemic infection
* Severe uncontrolled psychiatric illness
* Coagulopathy or anticoagulation therapy contraindicating surgery
* Pregnancy
* Previous extensive surgical interventions on the same site interfering with planned procedure
* Inability to comply with follow-up
* Any other condition that, in the opinion of the investigator, makes participation unsafe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Change in Pain (VAS Score) | Baseline, 10-12 days post-op, 3 months post-op
  Change in pain intensity measured using the visual analogue scale (0-10) to evaluate the clinical effect of surgical intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Nové Město Na Moravě, Nové Město na Moravě, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oaklander AL, Fields HL. Is reflex sympathetic dystrophy/complex regional pain syndrome type I a small-fiber neuropathy? Ann Neurol. 2009 Jun;65(6):629-38. doi: 10.1002/ana.21692. PMID 19557864
- [Background] Goebel A, Barker CH, Turner-Stokes L, et al. Complex regional pain syndrome in adults: UK guidelines for diagnosis, referral and management. Rheumatology (Oxford). 2018;57(8):1405-1436. PMID: 29648652
- [Background] Harden NR, Bruehl S, Perez RSGM, Birklein F, Marinus J, Maihofner C, Lubenow T, Buvanendran A, Mackey S, Graciosa J, Mogilevski M, Ramsden C, Chont M, Vatine JJ. Validation of proposed diagnostic criteria (the "Budapest Criteria") for Complex Regional Pain Syndrome. Pain. 2010 Aug;150(2):268-274. doi: 10.1016/j.pain.2010.04.030. Epub 2010 May 20. PMID 20493633